CLINICAL TRIAL: NCT02066350
Title: Assessment of Cardiovascular Risk Factors, Including Endothelial Function, After Restoration of Normoglycemia Following Single Pancreas Transplantation
Brief Title: Cardiovascular Risk Factors After Single Pancreas Transplantation
Acronym: Diamant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Trond Jenssen, MD, PhD, Professor of Medicine, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/1062; 2013047 (Other Grant/Funding Number: South-Eastern Norway Regional Health Authority)
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Type 1; Endothelial Dysfunction
Keywords: Diabetes type 1; Endothelial dysfunction; Pancreas transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single pancreas transplantation (Experimental): This is an explorative analysis to assess the impact of establishing normoglycemia in previously hyperglycemic patients, without using antidiabetic drugs, by investigating patients before and after single pancreas transplantation. Active patients on the waiting list for single pancreas transplantation will be investigated while on the waiting list and subsequently 8 weeks and 1 year after transplantation if they have a functioning pancreas graft. A control group of healthy volunteers (non-diabetic, non-transplanted), frequency-matched for age and gender with regards to the pancreas transplanted patients, will be investigated once.
  Interventions: Procedure: Single pancreas transplantation

INTERVENTIONS:
Procedure: Single pancreas transplantation

SUMMARY:
Patients accepted for the waiting list for single pancreas transplantation suffer from severe glucose instability with hyperglycemia due to diabetes type 1, but do not have significant diabetes-related complications. Pancreas transplantation restores normoglycemia in diabetes type 1 patients with unstable control of glycemia. Both hypo- and hyperglycemic events are abolished, and 70-80 % of the patients obtain satisfactory HbA1c levels (HbA1c 5.0-6.0 %) without the need of exogenous insulin. Endothelial dysfunction is considered as an early and potentially reversible stage in the atherosclerotic process. The endothelium is involved in homeostasis, leucocyte adhesion and vasomotor activity. Reduced endothelium-dependent vasodilation is associated with increments in cardiovascular risk factors, and endothelial dysfunction is a predictor for future cardiovascular disease. It has also been hypothesized that endothelial dysfunction may be involved in the impaired glycemic control by reducing the availability of glucose in peripheral muscles.Establishing normoglycemia by pancreas transplantation alone in previously diabetic type 1 patients has recently been shown to improve left ventricular ejection fraction, assessed by Doppler echocardiographic examination. In diabetic patients receiving a new pancreas it is possible to assess the effect of changing blood glucose excursions on cardiovascular risk factors, including endothelial function, without the use of antidiabetic drugs (exclude pleiotropic effects).

The primary objective of the present study is to assess if endothelial function (assessed by flow-mediated dilatation of arteria brachialis) is improved when hyperglycemia is reversed by single pancreas transplantation in patients with type 1 diabetes.

Secondary objectives are to investigate the changes in the following parameters by reversal of hyperglycemia by pancreas transplantation; Peripheral arterial tonometry, serum/plasma concentrations of endothelial dysfunction markers, blood pressure, lipid and lipoprotein concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes accepted for the waiting list for single pancreas transplantation
* Healthy volunteers (non-diabetic, non-transplanted)
* Over 18 years of age
* Signed informed consent

Exclusion Criteria:

* Non-functioning pancreas graft (defined as HbA1c ≥ 6.5 % with the need of insulin injections and fasting C-peptide concentration < 300 pmol/L).
* Active infection
* Active autoimmune disease other than diabetes
* Severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 1 year post-transplant
  This is an explorative analysis to assess the impact of establishing normoglycemia in previously hyperglycemic patients, without using antidiabetic drugs, by investigating patients before and after single pancreas transplantation. Active patients on the waiting list for single pancreas transplantation will be investigated while on the waiting list and subsequently 8 weeks and 1 year after transplantation if they have a functioning pancreas graft. Flow-mediated dilatation (FMD) of large vessels (arteria brachialis) will be assessed by measuring vessel diameter by ultrasound and the FMD of micro vessels in the finger tip will be assessed by Endo-PAT (PAT=Peripheral Arterial Tonus) following reactive hyperperfusion induced by occlusion of the artery by a sphygmomanometer cuff.

SECONDARY OUTCOMES:
Peripheral arterial tonometry | 1 year post-transplant
Changes in cardiac performance | 1 year post-transplant
  An echocardiographic examination will be performed to assess changes in cardiac performance, such as left ventricular ejection fraction
Pulse wave velocity (arterial stiffness) | 1 year post-transplant
  Pulse wave velocity, using a SphygmoCor device, measuring arterial stiffness will be performed in addition to pulse wave analysis evaluating the shape and amplitude of the aortic pulse wave.
Heart rate variability | 1 year post-transplant
  Heart rate variability will be assessed, using a Vagus device, analyzing short-term electrocardiogram recordings.
Plasma concentrations of endothelial dysfunction markers | 1 year post-transplant
  Fasting plasma samples (6 mL EDTA vacutainer) will be drawn for determination of relevant markers for endothelial dysfunction, such as von Willebrand factors (vWF) and vascular cell adhesion molecule-1 (VCAM-1).
Blood pressure | 1 year post-transplant
  Blood pressure will be measured seated after ten minutes rest by Dyna Map (Tuff.-Cuff, CAS Medical system Inc.) and the mean of the lower two out of three measurements will be used.
Lipid and lipoprotein concentrations | 1 year post-transplant
Bone mineral density and body composition | 1 year post-transplant
  Measurement of bone mineral density, using low dosage radiation (dual-energy X-ray absorptiometry (DEXA) scan) to assess the amount (grams) of mineral that are packed into a segment of bone. In addition a body composition (visceral fat, metabolic measurement) will be determined using the DEXA scan.
Glomerular filtration rate | 1 year post-transplant
  Renal function, defined as glomerular filtration rate, will be evaluated by measuring iohexol clearance. The concentration of iohexol (Omnipaque), a low dose non-ionic x-ray contrast medium of low osmolality, extensively used in clinical radiology and considered essentially free from side effects, will be measured 2 hours and 5 hours after iv injection of iohexol. Like other iodine-containing contrast media, it is completely eliminated from the body by excretion in the urine, thus it is an ideal marker for kidney function. It will be quantitated by chemical measurement based on the determination of iodine.
Oral glucose tolerance test | 1 year post-transplant
  Measurements of plasma glucose, C-peptide and serum insulin before, 30 and 120 minutes following an oral administration of 75 g glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Trond G Jenssen, Professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway